CLINICAL TRIAL: NCT01808326
Title: A Phase II, Open Label, Single Arm, Multicenter Study of Chlorambucil in Japanese Previously Untreated Patients With Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 116586
Record Dates: First submitted 2013-02-21; First posted 2013-03-11 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2015-06-22 (Estimated); Status verified 2015-04

CONDITIONS: Leukaemia, Lymphoblastic
MeSH Terms: conditions — Leukemia | interventions — Chlorambucil; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- chlorambucil (Experimental): chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 treatment cycles
  Interventions: Drug: chlorambucil, tablets

INTERVENTIONS:
Drug: chlorambucil, tablets — 2mg tablets, chlorambucil dose: 10mg/m2 PO at days 1-7 every 28 days; duration: minimum of 3 cycles until best response or maximum of 12 cycles

SUMMARY:
This study is an open-label, single arm, phase II study of chlorambucil in subjects with previously untreated CLL.

The primary objective is to evaluate the response to chlorambucil in Japanese subjects with previously untreated CLL.

Secondary objectives are to evaluate efficacy, safety and pharmacokinetics of chlorambucil in Japanese subjects.

DETAILED DESCRIPTION:
This study is an open-label, single arm, phase II study of chlorambucil in subjects with previously untreated CLL.

The primary objective is to evaluate the response to chlorambucil in Japanese subjects with previously untreated CLL.

Secondary objectives are to evaluate efficacy, safety and pharmacokinetics of chlorambucil in Japanese subjects.

Chlorambucil is an effective and well-tolerated chemotherapeutic agent currently approved for treatment of chronic lymphocytic leukemia (CLL) in the United States of America (US), European Union (EU) and other countries globally but not in Japan. Other more aggressive treatment options such as a combination of fludarabine (F) and cyclophosphamide are available, but are associated with significantly greater toxicities. The addition of ofatumumab to chlorambucil offers potentially a more effective therapy, with limited additional toxicity.

Study OMB110911 has been conducted mainly in the US and EU to evaluate progression-free survival (PFS) and overall response (OR) in subjects with previously untreated CLL with ofatumumab in combination with chlorambucil versus (vs.) chlorambucil monotherapy.

The objective of this study is to evaluate overall response of chlorambucil in Japanese subjects with previously untreated CLL.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL defined by:Circulating B lymphocytes ≥5,000 /μL AND Flow cytometry confirmation of immunophenotype with CD5, CD19, CD20, and CD23 prior to Visit 2.
* Considered inappropriate for fludarabine-based therapy.
* Active disease and indication for treatment based on the IWCLL updated NCI-WG guidelines defined by presenting at least any one of the following conditions: Evidence of progressive marrow failure as manifested by development or worsening of anemia and/or thrombocytopenia.

Massive (i.e. at least 6 cm below the left costal margin) or progressive or symptomatic splenomegaly.

Massive nodes (i.e. at least 10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.

Progressive lymphocytosis with an increase of more than 50% over a two month period or an lymphocyte doubling time of less than 6 months.

A minimum of any one of the following disease-related symptoms must be present: a) Unintentional weight loss ≥10% within the previous six months; b) Fevers >38.0°C for ≥ 2 weeks without evidence of infection; or c) Night sweats for more than 1 month without evidence of infection

* Not been previously treated for CLL (prior autoimmune hemolytic anemia treatment with corticosteroids permitted).
* ECOG Performance Status of 0-2.
* QTc <450 msec or QTc <480 msec for patients with bundle branch block The QTc is the QT interval corrected for heart rate according to either Bazett's formula (QTcB) or to Fridericia's formula (QTcF), machine or manual overread, for males and females. The specific formula that will be used in a protocol should be determined prior to initiation of the study, and the formula used to determine inclusion and discontinuation should be the same throughout the study.

The QTc should be based on single or averaged QTc values of triplicate electrocardiograms (ECGs) obtained over a brief recording period.

* Life expectancy of at least 6 months, in the opinion of the investigator.
* Age ≥ 20 years
* Signed written informed consent prior to performing any study-specific procedures (the results of other procedures predating the informed consent can be used).

Exclusion Criteria:

* Prior immuno- or chemotherapy for CLL or small lymphocytic lymphoma (SLL) with any agent except corticosteroids used to treat autoimmune hemolytic anemia.
* Previous autologous or allogeneic stem cell transplantation.
* Active autoimmune hemolytic anemia (AIHA) requiring corticosteroid therapy >100 mg/day equivalent to hydrocortisone, or chemotherapy.
* Known transformation of CLL (e.g. Richter).
* Known CNS involvement of CLL.
* Chronic or current active infectious disease requiring systemic antibiotics, antifungal, or antiviral treatment such as, but not limited to, chronic renal infection, chronic chest infection with bronchiectasis, tuberculosis and active Hepatitis C.
* Other past or current malignancy. Subjects who have been free of malignancy for at least 5 years, or have a history of completely resected non-melanoma skin cancer, or successfully treated in situ carcinoma are eligible.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months prior to screening, congestive heart failure, and arrhythmia requiring therapy, with the exception of extra systoles or minor conduction abnormalities.
* History of significant cerebrovascular disease or event with significant symptoms or sequelae.
* Glucocorticoid use, unless given in doses ≤ 100 mg/day hydrocortisone (or equivalent dose of other glucocorticoid) for <7 days for exacerbations other than CLL (e.g. asthma).
* Known HIV positive.
* Positive serology for Hepatitis B (HB) defined as a positive test for HBsAg. In addition, if negative for HBsAg but HBcAb and/or HBsAb positive, an HBV DNA test will be performed, and if positive the subject will be excluded.
* Screening laboratory values:

Creatinine >2.0 times upper normal limit (unless normal creatinine clearance). Total bilirubin > 2.0 times upper normal limit (unless due to Gilbert's syndrome).

Alanine aminotransferase (ALT) > 3.0 times upper normal limit.

* Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to Visit 1, whichever is longer, treatment with any anti-CD20 monoclonal antibody within 3 months of Visit 1, or participation in any other interventional clinical study.
* Known or suspected inability to comply with study protocol.
* Lactating women, women with a positive pregnancy test within 7 days prior to administration of the investigational product or women (of childbearing potential) as well as men with partners of childbearing potential, who are not willing to use adequate contraception from study start through one year following last treatment dose. Adequate contraception is defined as oral hormonal birth control, intrauterine device, and male partner sterilization (if male partner is sole partner for that subject) and the double barrier method (condom or occlusive cap plus spermicidal agent).

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-04; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Japan (5):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Fukuoka
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Tokyo

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study consisted of three phases: Screening Phase (within 6 weeks prior to Day 1), Treatment Phase (up to 48 weeks) and Follow-up Phase (up to 24 Weeks).
Pre-assignment Details: Participants with Chronic Lymphocytic Leukemia (CLL) were enrolled after blood sampling, physical examination, and Computed Tomography (CT) scan. The physical examination was performed <=14 days prior to Visit 2, CT scan performed within 6 weeks and the bone marrow examination within 6 weeks prior to Day 1.
Groups:
- Chlorambucil 10 mg/m^2: Participants with previously untreated chronic lymphocytic leukemia (CLL) received chlorambucil 10 milligram (mg)/meter squared (m^2) orally on Days 1-7 of every 28-day cycle for a minimum of 3 cycles until best response or a maximum of 12 cycles. After completion of the Treatment Phase (for participants in CR, PR or SD), survival and disease status assessment visits were performed 28 days after the first day of the last treatment cycle (Follow-up [FU] 1), 84 days, and 168 days after the day of FU 1 (FU 85 and FU 169, respectively). For participants experiencing disease progression during the Treatment Phase, the post progressive disease (PD) follow-up for safety assessments were performed 28 days after the first day of the last treatment cycle (PDFU 1). Subsequent follow-up was performed 84 and 168 days after the day of PDFU 1 (PDFU 85 and PDFU 169, respectively) to assess survival status, date of next CLL therapy, and type of therapy. In subsequent visits, the participant continued
Period: Overall Study
Arm/Group | Chlorambucil 10 mg/m^2
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (7.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian - Japanese Heritage | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Best Response of Either Complete Remission (CR), Nodular Partial Remission (nPR), Complete Remission-incomplete (CRi) or Partial Remission (PR), as Assessed by the Investigator, IRC and IRC With CT
Description: According to the criteria based on the 2008 revision of the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) of the National Cancer Institute-Sponsored Working Group Guidelines (NCI-WG), participants with complete remission (CR), nodular partial remission (nPR), complete remission-incomplete (CRi) and partial remission (PR) were classified as responders, while stable disease (SD) and progressive disease (PD) were classified as non-responders. Participants with unknown or missing responses were considered as non-responders. Assessment was completed by the Investigator, Independent Review Committee (IRC), and IRC with Computed Tomography (CT).
Time Frame: From the start of treatment until disease progression or death (up to Week 61.1)
Population: All Subjects Population: all participants who received at least one dose of investigational product.
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  IRC with CT Assessed | 3
  IRC Assessed | 5
  Investigator-Assessed | 5

2. Secondary Outcome: Number of Participants With the Best Overall Response (OR), as Assessed by the Investigator, IRC and IRC With CT
Description: OR is defined as the number of participants achieving either a confirmed CR or PR. Assessment was completed by the Investigator, IRC, and IRC with CT. CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM.
Time Frame: From the start of treatment until disease progression or death (up to Week 61.1)
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  Investigator-Assessed, CR | 0
  Investigator-Assessed, CRi | 0
  Investigator-Assessed, nPR | 0
  Investigator-Assessed, PR | 5
  Investigator-Assessed, Responders | 5
  IRC Assessed, CR | 0
  IRC Assessed, CRi | 0
  IRC Assessed, nPR | 0
  IRC Assessed, PR | 5
  IRC Assessed, Responders | 5
  IRC with CT Assessed, CR | 0
  IRC with CT Assessed, CRi | 0
  IRC with CT Assessed, nPR | 0
  IRC with CT Assessed, PR | 3
  IRC with CT Assessed, Responders | 3

3. Secondary Outcome: Progression Free Survival (PFS), as Assessed by the Investigator and the IRC
Description: Progression-free survival (PFS) is defined as the time from the start of treatment of investigational product until the first documented sign of PD or death due to any cause. PD requires at least one of the following: lymphadenopathy, appearance of any new lesion such as enlargerd lymph nodes (>1.5 cm) spleen or liver or other infiltrates or an increase by 50% or more in the greatest diameter of any previous site; an increase by 50% or more in the previously noted enlargement of the liver or spleen, an increase by 50% or more in the numbers of blood lymphocytes with at least 5000 lymphocytes per microliter, transformation to a more aggressive histology, or occurrence of cytopenia attributable to chronic lymphocytic leukaemia. Par. who were alive and had not progressed at the time of analysis or if a progression event or death occurred after extensive lost-to-follow-up time or if new anti-cancer therapy was started were censored at the date of the last visit with adequate assessment.
Time Frame: From the start of treatment until disease progression or death (up to Week 61.1)
Population: All Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Weeks
  IRC Assessed | NA [NA to NA] — No PFS could be determined because no progression or death was observed in the participants up to follow up 28 weeks after the final day of the last treatment, and all participants were censored for analysis.
  Investigator Assessed | NA [NA to NA] — No PFS could be determined because no progression or death was observed in the participants up to follow up 28 weeks after the final day of the last treatment, and all participants were censored for analysis.

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as time from the start of treatment until death due to any cause. Participants who had not died were censored at the date of last contact.
Time Frame: From the start of treatment until death (up to Week 61.1)
Population: All Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Weeks | NA [NA to NA] — All 5 participants were alive at the time of the last follow-up and thus were censored for the analysis

5. Secondary Outcome: Time to Response, as Assessed by the IRC
Description: Time to response is defined as time from the start of treatment until the first response (CR/PR). Time to Response analyses was restricted to the subgroup of the population who experienced an overall response (CR/ nPR/CRi/PR) during the study. CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM.
Time Frame: From the start of treatment until the first response (CR/PR) (up to Week 61.1)
Population: All Subjects Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the All Subjects Population.
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Weeks | 4.1 [4.1 to 25.0]

6. Secondary Outcome: Duration of Response, as Assessed by the IRC
Description: Duration of response is defined as the time from the initial response (CR or PR) until progression or death. CR (all the criteria at least 2 months after last treatment): no lymphadenopathy (Ly) > 1.5 cm/ hepatomegaly/ splenomegaly/ constitutional symptoms; neutrophils >1500 per microliter (µL), platelets (PL) >100,000/µL, hemoglobin (Hb) >11 grams/deciliter (g/dL), lymphocytes (LC) <4000/µL, bone marrow (BM) sample must be normocellular for age, <30% LC, no lymphoid nodule. CRi: CR criteria, persistent anemia/thrombocytopenia/neutropenia unrelated to CLL but related to drug toxicity. PR: >=50% decrease in LC, Ly, size of liver and spleen and at least one of the following results: PL >100,000/µL or 50% improvement over Baseline (BL), Hb >11 g/dL or 50% improvement over BL. nPR: persistent nodules BM.
Time Frame: From the initial response (CR/PR) until disease progression or death (up to Week 61.1)
Population: All Subjects Population
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Weeks | NA [NA to NA] — The duration of response could not be assessed because no progression was observed in any of 5 participants up to Week 72

7. Secondary Outcome: Time to Next Chronic Lymphocytic Leukemia (CLL) Therapy
Description: Time to next CLL therapy is defined as the time from start of treatment until the first administration of the next CLL treatment other than chlorambucil administrations scheduled in this study. Time to next CLL therapy was restricted to the subgroup of the population who receive a next CLL therapy after experiencing disease progression.
Time Frame: From the start of treatment until the first administration of the next CLL treatment (up to Week 61.1)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Weeks | NA [NA to NA] — No data were available because no participants received the next CLL therapy

8. Secondary Outcome: Number of Participants With Improvement in Eastern Cooperative Oncology Group (ECOG) Performance Status (PS)
Description: ECOG PS is a scale to assess disease progression, extent to which disease affects the daily living abilities and determines appropriate treatment and prognosis. It is scored on a scale of 0 to 5 as, 0 (fully active), 1 (restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature), 2 (ambulatory and capable of all self cares but unable to carry out any work activities, Up and about > 50% of waking hours), 3 (capable of only limited self cares, confined to bed or chair > 50% of waking hours), 4 (completely disabled, cannot carry on any self cares, totally confined to bed or chair), 5 (death). Improvement is defined as decrease from baseline by at least one step on the ECOG performance status scale (yes/no). Baseline was last pre-dose assessment performed on Cycle 1 Day 1(C1 D1). When C1 D1 was missing, the last assessment performed prior to pre-dose C1 D1 was used. It was performed on Day 1 of each cycle and follow-up (FU).
Time Frame: Baseline, Cycle (C) 2-Day (D) 29, C3-D57, C4-D85, C5-D113, C6-D141, C7-D169, C8-D197, C9-D225, FU 1- PDFU 1, FU 85-PDFU 85, and FU 169-PDFU 169
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  Cycle 2-Day 29, Improved, n=5 | 0
  Cycle 2-Day 29, No Change, n=5 | 5
  Cycle 2-Day 29, Deteriorated, n=5 | 0
  Cycle 3-Day 57, Improved, n=4 | 0
  Cycle 3-Day 57, No Change, n=4 | 4
  Cycle 3-Day 57, Deteriorated, n=4 | 0
  Cycle 4-Day 85, Improved, n=4 | 0
  Cycle 4-Day 85, No Change, n=4 | 4
  Cycle 4-Day 85, Deteriorated, n=4 | 0
  Cycle 5-Day 113, Improved, n=4 | 0
  Cycle 5-Day 113, No Change, n=4 | 4
  Cycle 5-Day 113, Deteriorated, n=4 | 0
  Cycle 6-Day 141, Improved, n=4 | 1
  Cycle 6-Day 141, No Change, n=4 | 3
  Cycle 6-Day 141, Deteriorated, n=4 | 0
  Cycle 7-Day 169, Improved, n=1 | 0
  Cycle 7-Day 169, No Change, n=1 | 1
  Cycle 7-Day 169, Deteriorated, n=1 | 0
  Cycle 8-Day 197, Improved, n=1 | 0
  Cycle 8-Day 197, No Change, n=1 | 1
  Cycle 8-Day 197, Deteriorated, n=1 | 0
  Cycle 9-Day 225, Improved, n=1 | 0
  Cycle 9-Day225, No Change, n=1 | 1
  Cycle 9-Day 225, Deteriorated, n=1 | 0
  FU 1-PDFU 1, Improved, n=5 | 0
  FU 1-PDFU 1, No Change, n=5 | 5
  FU 1-PDFU 1, Deteriorated, n=5 | 0
  FU 85-PDFU 85, Improved, n=5 | 1
  FU 85-PDFU 85, No Change, n=5 | 4
  FU 85-PDFU 85, Deteriorated, n=5 | 0
  FU 169-PDFU 169, Improved, n=5 | 1
  FU 169-PDFU 169, No Change, n=5 | 4
  FU 169-PDFU 169, Deteriorated, n=5 | 0

9. Secondary Outcome: Number of Participants With no B-symptoms and With at Least One B-symptom Over Time
Description: The number of participants with no B-symptoms (no night sweat, no weight loss, no fever and no extreme fatigue) and the number of participants with at least one of the B-symptoms are summarized by assessment time. The presence of the B-symptoms was assessed at Baseline, Day 1 of each treatment cycle and follow-up (FU). Baseline was the last pre-dose assessment performed at C1 D1.
Time Frame: Baseline, C2-D29, C3-D57, C4-D85, C5-D113, C6-D141, C7-D169, C8-D197, C9-D225, FU 1-PDFU 1, FU 85-PDFU 85, and FU 169-PDFU 169
Population: as for outcome 5
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  Baseline, With no B-symptom, n=5 | 3
  Baseline, With at least one B-symptom, n=5 | 2
  Cycle 2-Day 29, With no B-symptom , n=5 | 4
  Cycle 2-Day 29, With at least one B-symptom, n=5 | 1
  Cycle 3-Day 57, With no B-symptom, n=4 | 4
  Cycle 3-Day 57, With at least one B-symptom, n=4 | 0
  Cycle 4-Day 85, With no B-symptom, n=4 | 4
  Cycle 4-Day 85, With at least one B-symptom, n=4 | 0
  Cycle 5-Day 113, With no B-symptom, n=4 | 4
  Cycle 5-Day 113, With at least one B-symptom, n=4 | 0
  Cycle 6-Day 141, With no B-symptom, n=4 | 4
  Cycle 6-Day 141, With at least one B-symptom, n=4 | 0
  Cycle 7-Day 169, With no B-symptom, n=1 | 1
  Cycle 7-Day 169, With at least one B-symptom, n=1 | 0
  Cycle 8-Day 197, With no B-symptom, n=1 | 1
  Cycle 8-Day 197, With at least one B-symptom, n=1 | 0
  Cycle 9-Day 225, With no B-symptom, n=1 | 1
  Cycle 9-Day 225,With at least one B-symptom, n=1 | 0
  FU 1-PDFU 1,With no B-symptom, n=5 | 5
  FU 1-PDFU 1,With at least one B-symptom, n=5 | 0
  FU 85-PDFU 85,With no B-symptom ,n=5 | 5
  FU 85-PDFU 85,With at least one B-symptom, n=5 | 0
  FU 169-PDFU 169, With no B-symptom, n=5 | 5
  FU 169-PDFU 169, With at least one B-symptom, n=5 | 0

10. Secondary Outcome: Number of Participants With Any Adverse Events (AE) or Serious Adverse Events (SAE)
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that, at any dose results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, is a congenital anomaly/birth defect or is associated with protocol specified liver injury and impaired liver function or is any protocol specific AEs.
Time Frame: From the start of treatment up to Week 61.1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  Any AE | 5
  Any SAE | 1

11. Secondary Outcome: Number of Participants With Adverse Events by the Indicated Maximum Toxicity Grade
Description: An AE is defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product whether or not considered related to the medicinal product. Non-hematologic AEs were graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 (NCI CTCAE V4.03): Grade 0, none; Grade 1, mild; Grade 2, moderate; Grade 3, severe or medically significant; Grade 4, life-threatening consequences; Grade 5, death related to AE
Time Frame: From the start of treatment up to Week 61.1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  Grade 1 | 0
  Grade 2 | 2
  Grade 3 | 3
  Grade 4 | 0
  Grade 5 | 0

12. Secondary Outcome: Number of Participants With at Least One Grade 3/Grade 4 Adverse Event of Infection or Myelosuppression (Anemia, Neutropenia, and Thrombocytopenia)
Description: Number of participants with a Grade 3 or Grade 4 adverse event of infection or myelosuppression (anemia, neutropenia, and thrombocytopenia) are presented. Myelosuppression is defined as the decrease in the ability of the bone marrow to produce blood cells. AEs were graded according to NCI common terminology criteria for adverse events (CTCAE) grade, version 3.0 (1, mild; 2, moderate; 3, severe; 4, life-threatening/disabling; 5, death).
Time Frame: From the start of treatment up to Week 61.1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants
  Infection, Grade 3 | 0
  Infection, Grade 4 | 0
  Myelosuppression, Grade 3 | 3
  Myelosuppression, Grade 4 | 0

13. Secondary Outcome: Change From Baseline in the Immunoglobulin(Ig) Antibodies IgA, IgG, and IgM
Description: Immunoglobulins, or antibodies, are large proteins used by the immune system to identify and neutralize foreign particles such as bacteria and viruses. Their normal blood levels indicate proper immune status. Low levels indicate immuno-suppression. IgA, IgG, and IgM were measured in the blood samples of the participants.Peripheral samples were collected for the analysis of IgA, IgG, and IgM at Baseline and 28 days after Day 1 of the last treatment cycle (FU 1-PDFU 1) for all participants, and 168 days after day of FU 1-PDFU 1 for participants with CR, PR, and SD. Baseline was the last pre-dose assessment performed on Cycle 1-Day 1. The the last assessment performed prior to pre-dose Cycle 1-Day 1 was used if Cycle 1-Day 1 was missing. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline, FU 1-PDFU 1, FU 85-PDFU 85, and FU 169-PDFU 169
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Grams per liter
  IgA, FU 1-PDFU 1, n=5 | -0.092 (0.2792)
  IgA, FU 169-PDFU 169, n=4 | -0.053 (0.2185)
  IgG, FU 1-PDFU 1, n=5 | -0.446 (1.2509)
  IgG, FU 169-PDFU 169, n=4 | 0.340 (0.8328)
  IgM, FU 1-PDFU 1, n=4 | -0.068 (0.3402)
  IgM, FU 169-PDFU 169, n=3 | 0.113 (0.1185)

14. Secondary Outcome: Number of Participants With Positive Minimal Residual Disease (MRD)
Description: MRD refers to the small number of leukemic cells that remain in the participant during treatment or after treatment at the time the participant achieved a confirmed CR and in whom bone marrow test was performed. A bone marrow sample was examined by flow cytometry (Cluster of differentiation [CD]5, CD19, CD20, and CD23). MRD positive is defined as more than one CLL cell per 10000 leukocytes.
Time Frame: From the start of treatment up to Week 61.1
Population: All Subjects Population
Measure: Number; unit: Participants
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Participants | 1

15. Secondary Outcome: Expression of Beta 2 Microglobulin
Description: Blood samples were collected at the Baseline (Day 1 of Cycle 1) visit for prognostic biomarker Beta 2 microglobulin measurements.
Time Frame: Baseline (Cycle 1 Day 1)
Population: All Subjects Population
Measure: Mean (Standard Deviation); unit: Nanomoles per Liter
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Nanomoles per Liter | 263.3906 (25.82599)

16. Secondary Outcome: Expression of Complement CH50
Description: Peripheral samples were collected for the analysis of complement CH50 at Baseline (Day 1 of Cycle 1) and after completion of Cycle 4 (Day 85).
Time Frame: Baseline, Cycle 1-Day 1, and Cycle 4-Day 85
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Kilounit /Liter
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Kilounit /Liter
  Cycle 1-Day 1, n=4 | 45.48 (3.037)
  Cycle 4-Day 85, n=4 | 40.08 (10.942)

17. Secondary Outcome: Maximum Serum Concentration (Cmax), and Minimum Serum Concentration (Cmin) for Chlorambucil
Description: Blood samples for pharmacokinetic (PK) analysis of chlorambucil were collected on Day 1 and Day 4 in Cycle 1, and on Day 1 in Cycle 3. In each sampling, blood samples (2 milliliter [mL]/sample) were collected at pre-dose, and 15 minute (min), 30 min, 1 hour (hr), 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. Maximum serum concentration (Cmax), minimum serum concentration (Cmin) were determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 1
Population: PK Population: all participants who received at least one dose of investigational product and for whom PK data was collected. Only those participants with non-missing values available at the specified time points were analyzed (represented by n=X in the category titles).
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Nanograms per milliliter
  Cmax, Cycle 1-Day 1, n=5 | 746.846 [499.393 to 1116.913]
  Cmax, Cycle 1-Day 4, n=4 | 884.046 [679.823 to 1149.621]
  Cmax, Cycle 3-Day 57, n=4 | 691.960 [553.342 to 865.303]
  Cmin, Cycle 1-Day 4, n=5 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points.
  Cmin, Cycle 3-Day 57, n=4 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points.

18. Secondary Outcome: Area Under the Serum Concentration-time (AUC) for Chlorambucil
Description: Blood samples for PK analysis of chlorambucil were collected on Day 1 and Day 4 in Cycle 1, and on Day 57 in Cycle 3. In each sampling, blood samples (2 mL/sample) were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. AUC from time zero up to a definite time t (AUC[0-t]), AUC from time zero up to infinity (AUC[0-inf]), AUC from time zero up to 6 hours post dose (AUC[0-6]), AUC from time zero up to 24 hours post dose (AUC[0-24]) were determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: PK Population. Only those participants available at the specified time points were analyzed (represented by n=X in the category titles). Different participants may have been analyzed at different time points, so the overall number of participants analyzed reflects everyone in the PK Population.
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*nanogram/ milliliter/milligram
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Hour*nanogram/ milliliter/milligram
  AUC(0-t), Cycle 1-Day 1, n=5 | 1207.8510 [890.7718 to 1637.7978]
  AUC(0-t),Cycle 1-Day 4, n=4 | 1391.5506 [1078.6087 to 1795.2878]
  AUC(0-t), Cycle 3-Day 57, n=4 | 1274.2668 [1043.5229 to 1556.0327]
  AUC(0-inf), Cycle 1-Day 1, n=5 | 1230.8109 [910.1764 to 1664.3978]
  AUC(0-inf), Cycle 1-Day 4, n=4 | 1408.1764 [1094.5401 to 1811.6841]
  AUC(0-inf), Cycle 3-Day 57, n=4 | 1354.2258 [960.1552 to 1910.0323]
  AUC(0-24), Cycle 1-Day 1, n=5 | 1230.6335 [910.0130 to 1664.2168]
  AUC(0-24), Cycle 1-Day 4, n=4 | 1408.1363 [1094.5040 to 1811.6406]
  AUC(0-24), Cycle 3-Day 57, n=4 | 1334.2607 [990.8919 to 1796.6153]
  AUC(0-6), Cycle 1-Day 1, n=5 | 1183.4581 [869.4781 to 1610.8205]
  AUC(0-6), Cycle 1-Day 4, n=4 | 1375.8404 [1081.1272 to 1750.8917]
  AUC(0-6), Cycle 3-Day 57, n=4 | 1246.9176 [1056.4256 to 1471.7587]

19. Secondary Outcome: Elimination Half-life (t1/2) for Chlorambucil
Description: Blood samples for pharmacokinetic (PK) analysis of chlorambucil were collected on Day 1 and Day 4 in Cycle 1, and on Day 57 in Cycle 3. In each sampling, blood samples (2 mL/sample) were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. Elimination half-life (t1/2) was determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Hour
  t1/2, Cycle 1-Day 1 , n=5 | 1.3488 [1.0090 to 1.8030]
  t1/2, Cycle 1-Day 4, n=5 | 1.3211 [0.9035 to 1.9316]
  t1/2, Cycle 3-Day 57, n=4 | 1.6979 [0.4245 to 6.7918]

20. Secondary Outcome: Time of Maximum Serum Concentration (Tmax) for Chlorambucil
Description: Blood samples for pharmacokinetic (PK) analysis of chlorambucil were collected on Day 1 and Day 4 in Cycle 1, and on Day 57 in Cycle 3. In each sampling, blood samples (2 mL/sample) were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. Time of maximum serum concentration (tmax) was determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Hour
  tmax, Cycle 1-Day 1, n=5 | 1.000 [0.95 to 1.50]
  tmax, Cycle 1-Day 4, n=4 | 0.725 [0.48 to 1.50]
  tmax, Cycle 3-Day 57, n=4 | 0.975 [0.50 to 1.48]

21. Secondary Outcome: Maximum Serum Concentration (Cmax), and Minimum Serum Concentration (Cmin) for Phenyl Acetic Acid Mustard
Description: Blood samples for pharmacokinetic (PK) analysis of chlorambucil and its metabolite phenyl acetic acid mustard were collected on Day 1 and Day 4 in Cycle 1, and on Day 1 in Cycle 3. In each sampling, blood samples (2 milliliter [mL]/sample) were collected at pre-dose, and 15 minute (min), 30 min, 1 hour (hr), 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. Maximum serum concentration (Cmax), minimum serum concentration (Cmin) were determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 1
Population: as for outcome 17
Measure: Geometric Mean (95% Confidence Interval); unit: Nanograms per milliliter
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Nanograms per milliliter
  Cmax, Cycle 1-Day 1, n=5 | 502.942 [418.135 to 604.949]
  Cmax, Cycle 1-Day 4, n=4 | 516.310 [406.414 to 655.923]
  Cmax, Cycle 3-Day 57, n=4 | 417.660 [345.801 to 504.451]
  Cmin, Cycle 1-Day 4, n=5 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points
  Cmin, Cycle 3-Day 57, n=4 | NA [NA to NA] — The Cmin value was non quantifiable (NQ) for all time points

22. Secondary Outcome: Area Under the Serum Concentration-time (AUC) for Phenyl Acetic Acid Mustard
Description: Blood samples for PK analysis of chlorambucil and its metabolite phenyl acetic acid mustard were collected on Day 1 and Day 4 in Cycle 1, and on Day 57 in Cycle 3. In each sampling, blood samples (2 mL/sample) were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. AUC from time zero up to a definite time t (AUC[0-t]), AUC from time zero up to infinity (AUC[0-inf]), AUC from time zero up to 6 hours post dose (AUC[0-6]), AUC from time zero up to 24 hours post dose (AUC[0-24]) were determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: Hour*nanogram/ milliliter/milligram
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Hour*nanogram/ milliliter/milligram
  AUC(0-t), Cycle 1-Day 1, n=5 | 1890.7202 [1657.6433 to 2156.5694]
  AUC(0-t),Cycle 1-Day 4, n=4 | 1902.4232 [1474.2957 to 2454.8766]
  AUC(0-t), Cycle 3-Day 57, n=4 | 1839.8498 [1375.6347 to 2460.7168]
  AUC(0-inf), Cycle 1-Day 1, n=5 | 2015.0708 [1783.4844 to 2276.7288]
  AUC(0-inf), Cycle 1-Day 4, n=4 | 2011.2434 [1521.8953 to 2657.9357]
  AUC(0-inf), Cycle 3-Day 57, n=4 | 2012.4576 [1422.5732 to 2846.9435]
  AUC(0-24), Cycle 1-Day 1, n=5 | 2013.1533 [1781.2371 to 2275.2649]
  AUC(0-24), Cycle 1-Day 4, n=4 | 2008.6155 [1521.3369 to 2651.9676]
  AUC(0-24), Cycle 3-Day 57, n=4 | 2007.1545 [1422.7652 to 2831.5771]
  AUC(0-6), Cycle 1-Day 1, n=5 | 1568.5579 [1339.5928 to 1836.6580]
  AUC(0-6), Cycle 1-Day 4, n=4 | 1647.7794 [1332.9712 to 2036.9359]
  AUC(0-6), Cycle 3-Day 57, n=4 | 1519.3633 [1215.2713 to 1899.5468]

23. Secondary Outcome: Elimination Half-life (t1/2) for Phenyl Acetic Acid Mustard
Description: Blood samples for pharmacokinetic (PK) analysis of chlorambucil and its metabolite phenyl acetic acid mustard were collected on Day 1 and Day 4 in Cycle 1, and on Day 57 in Cycle 3. In each sampling, blood samples (2 mL/sample) were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. Elimination half-life (t1/2) was determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 18
Measure: Geometric Mean (95% Confidence Interval); unit: Hour
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Hour
  t1/2, Cycle 1-Day 1 , n=5 | 2.0929 [1.7061 to 2.5674]
  t1/2, Cycle 1-Day 4, n=5 | 2.1846 [1.7179 to 2.7782]
  t1/2, Cycle 3-Day 57, n=4 | 2.3495 [1.4906 to 3.7031]

24. Secondary Outcome: Time of Maximum Serum Concentration (Tmax) for Phenyl Acetic Acid Mustard
Description: Blood samples for pharmacokinetic (PK) analysis of chlorambucil and its metabolite phenyl acetic acid mustard were collected on Day 1 and Day 4 in Cycle 1, and on Day 57 in Cycle 3. In each sampling, blood samples (2 mL/sample) were collected at pre-dose, and 15 min, 30 min, 1 hr, 1.5 hr, 2 hr, 3 hr, 4 hr, 6 hr, 8 hr, and 10 hr post dosing. Time of maximum serum concentration (tmax) was determined. Between participants coefficient of variation (%CVb) was calculated according to the following methods: Transformed Data : 100 * (square root of the exponential [standard deviation of loge-transformed ]2-1).
Time Frame: Cycle 1-Day 1, Cycle 1-Day 4, and Cycle 3-Day 57
Population: as for outcome 18
Measure: Median (Full Range); unit: Hour
Arm/Group | Chlorambucil 10 mg/m^2
Number analyzed (Participants) | 5
Hour
  tmax, Cycle 1-Day 1, n=5 | 1.970 [1.50 to 2.00]
  tmax, Cycle 1-Day 4, n=4 | 1.490 [1.47 to 2.00]
  tmax, Cycle 3-Day 57, n=4 | 1.730 [1.47 to 2.00]

ADVERSE EVENTS:
Time Frame: On-therapy serious adverse events (SAEs) and non-serious adverse events (AEs) were collected from the start of study treatment and until the follow-up contact (up to Week 61.1.
Description: On-therapy SAEs and non-serious AEs are reported for members of the All Subjects Population, comprised of all participants who received at least one dose of investigational product.
Arm/Group | Chlorambucil 10 mg/m^2
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorambucil 10 mg/m^2 (N=5)
Herpes zoster (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Chlorambucil 10 mg/m^2 (N=5)
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Neutropenia (Blood and lymphatic system disorders) | 4
Anaemia (Blood and lymphatic system disorders) | 2
White blood cell count decreased (Investigations) | 4
Aspartate aminotransferase increased (Investigations) | 2
Blood lactate dehydrogenase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 2
Alanine aminotransferase increased (Investigations) | 1
Blood alkaline phosphatase increased (Investigations) | 1
Haemoglobin decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Nausea (Gastrointestinal disorders) | 2
Abdominal discomfort (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Nasopharyngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Hypersensitivity (Immune system disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.